CLINICAL TRIAL: NCT03366922
Title: EVALUATION OF THE EFFECT OF ARTEMISIA ANNUA AND MORINGA OLEIFERA ON IMMUNOLOGICAL RESPONSE IN HAART HIV PATIENTS at MRRH
Brief Title: Evaluation of Artemisia Annua and Moringa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mbarara University of Science and Technology (Other)
Collaborators: ANAMED (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27/05-17
Record Dates: First submitted 2017-11-20; First posted 2017-12-08 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Participants will be stratified according to baseline CD4 levels: 350 - 250, 249 - 150, below 149. Computer generated numbers will be used to assign selected participants into study groups using simple randomization method to either control group with HAART only, or HAART with Artemisia annua group or HAART with Artemisia annua and Moringa oleifera group of 1:1:1.
Who Masked: Participant, Care Provider
Masking Description: * Two research assistants will be recruited and trained as observers and data collectors to increase accuracy and consistency in documenting the needed data. They will be assisted by the HIV clinic staff and these research assistants will be blinded to the hypotheses of this study to minimize observer bias and facilitate participant randomization. Senior clinician at the HIV clinic will supervise the trial and administration of treatments for HAART patients attending at the MRRH clinic.
  * To endure blinding, a study nurse will randomize and interview the participants and or draw blood whenever necessary. Study phlebotomist will draw blood and deliver it to the respective laboratory with codes masking the arm in which that patient is randomized. Independent laboratory technicians will run the tests at Epicenter and MUST research Labs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (Active Comparator): Participants will be on routine HAART only. No Artemisia Annua, Moringa oleifera will be given.
  Interventions: Dietary Supplement: Artemisia Annua, Moringa oleifera
- Intervention Arm 1 (Experimental): Participants will be given HAART and Artemisia annua leaf powder 4 g per day. They will only receive Artemisia Annua, Moringa oleifera will not be given.
  Interventions: Dietary Supplement: Artemisia Annua, Moringa oleifera
- Intervention Arm 2 (Experimental): Participants will be given HAART with Artemisia annua leaf powder of 4 grams per day and Moringa oleifera leaf powder of 10 grams per day. Both Artemisia Annua, Moringa oleifera will be given.
  Interventions: Dietary Supplement: Artemisia Annua, Moringa oleifera

INTERVENTIONS:
Dietary Supplement: Artemisia Annua, Moringa oleifera — As described above

SUMMARY:
Introduction Artemisia annua L is a medicinal plant traditionally used for treatment of malaria and other diseases in China. The extract of leaves of the plant has been demonstrated in-vitro to have potent anti HIV effects and in vivo to improve levels of lymphocytes in laboratory animals. Effect on lymphocyte stimulation has also been observed in non HIV persons taking the leaves of the plant as a tea for malaria prophylaxis in Uganda.

Objective To determine the effect of A.annua L and Moringa oleifera leaf powder on CD4 cell count and other immunological indices in HAART HIV patients.

Materials and Methods In this study Artemisia annua leaf powder and Moringa leaf powder will be investigated. The study will be a three arm randomized Phase II study involving adult patients with HIV-infection on HAART with CD4 below 350. The CD4 cell count, and other immunological indices in patients receiving HAART will be compared with those patients receiving additionally Artemisia annua powder with Moringa oleifera powder or Artemisia annua powder alone. The study will be conducted at the HIV clinic in Mbarara Regional Referral Hospital while laboratory tests will be done at Mbarara University of Science and Technology clinical and pharmaceutical sciences laboratories.

Expected outcome The primary outcome will be change in mean (Median) CD 4 cell count. Secondary outcomes will be mean (or median) changes, viral load, complete blood count and other HIV associated immunological indices , Performance status and incidence of adverse effects like nausea, diarrhoea, weight gain and or loss.

Expected benefits Adequate immunological recovery is one of the desired outcomes in HIV care. HAART combinations do not directly aid immunological recovery and some patients fail to have adequate immunological recovery despite adequate suppression of viral load. There are many patients using herbal supplements but there is limited scientific clinical evidence on the benefit of these supplements in HAART patients.

DETAILED DESCRIPTION:
HIV still remains a major public health burden in Uganda and Africa as a whole. It is estimated that about 36.9 million persons are infected worldwide with majority being in Africa. While most HIV persons in Uganda initiate HAART late sometimes with CD4 cell count below 350, making their immunological recovery very poor and putting them at higher risk of opportunistic infections, there are no established medicines for enhancement of immune responses.

Indeed a number of medicinal plants are reported to have anti-HIV effects and immune enhancement effect in vitro, however few to none have had their potential demonstrated in a controlled clinical study. This study will investigate A.annua supplemented with Moringa oleifera. Artemisia annua medicinal plant has been demonstrated to have immunological effects in laboratory studies as well as anti-HIV effects in vitro (Lubbe et al., 2012). Moringa oleifera has been reported to be used in up to 80% of HIV patients in Africa (Lubinga et al., 2012) and thus will be investigated as a nutritional supplement. Although there is improved access to testing and hence timely diagnosis for HIV with increased roll out of anti-retroviral therapy, many patients in resource limited settings still initiate HAART when the HIV-infection is in advanced stage. Initiation of HAART in patients with advanced HIV-infection has previously been associated with sub-optimal immunological recovery (Reda et al., 2012). In addition, in Uganda many HIV patients are reported to use herbal medicines in addition to HAART, including Aloe vera, Vernonia amygdalina and Moringa oleifera. (Lubinga et al., 2012). The challenge is that the clinical benefits of most of these herbal medicines remain unknown as well as their potential interactions with HAART. Artemisia annua powder which has been shown in vitro to have anti-HIV effects and in vivo to cause increase in monocytes and lymphocytes level (Lubbe et al., 2012; Ndhlala et al., 2016) is used by some HIV patients in Uganda claiming to improve their quality of life (Lubinga et al., 2012). However there are no data from controlled studies to prove these claims and thus enable adoption or rejection of Artemisia annua powder and Moringa oleifera as an adjunct to HIV treatment. Proof of beneficial effects of a given herbal remedy would provide an alternative to use of unproven herbal products as it is the case currently. Artemisia annua medicinal plant has been demonstrated to have immunological effects in laboratory studies as well as anti-HIV effects in vitro (Lubbe et al., 2012). Has a short plasma half-life. When given orally or rectally, dihydroartemisinin was safe and showed higher bioavailability in humans than artemisinin in an early pharmacokinetic study by Zhao et al (1993). The Cmax, Tmax, and T1/2 for orally delivered dihydroartemisinin were 0.13-0.71 mg/L, 1.33 h, approximately 1.6 h, respectively; for pure artemisinin they were 0.09 mg/L, 1.5 h, and 2.27 h, respectively. Alin et al (1996) compared orally delivered artemisinin and artemisinin-mefloquine combination therapy for treatment of P. falciparum malaria. Infected and uninfected patients had similar pharmacokinetic parameters. After a single dose, bioavailability of artemisinin was not altered. In the Ilet et al(2005) review of pharmacokinetic parameters of artemisinin and its derivatives, oral pure artemisinin doses ranged from about 6-11 mg kg/L in healthy subjects and Cmax was 0.15-0.39 mg/L. Dose seemed to have no major effect. An earlier study by Ashton et al (1998)compared increasing artemisinin doses of 250, 500, and 1000 mg per person and both Cmax and T1/2 showed dose-dependent increases of 0.21, 0.45, and 0.79 mg/L, and 1.38, 2.0, and 2.8 h, respectively, but Tmax remained relatively constant at 2.3-2.8 h. et al., (2011; 2012) has also found Artemisia tea at 2.5g dried leaves per adult infusion dose with 55-100mg artemisinin/L safe. Other pharmacokinetic studies have been duly added in the background section and show that artemisinin delivered by oral consumption of Artemisia annua dried leaves or encapsulated dried leaves of Artemisia Annua are generally safe (Weather et al., 2014; Elfawal et al., 2015; Desroslera and Weathers, 2016).

Moringa oleifera on the other hand has been reported to be used as a nutritional supplement and management of HIV infections in up to 80% of HIV patients in Africa (Monera et al., 2008; Lubinga et al., 2012; Popoola et al., 2013; Ndhlala et al., 2016; Roelofsen et al., 2017). Asare and colleagues (2012) also confirmed that intake of Moringa Oleifera is very safe at levels ≤ 1000 mg/kg b.wt. Monera and colleagues have also found out in a cross-over study that Co administration of Moringa oleifera Lam. leaf powder at the traditional dose did not alter the steady state pharmacokinetics of nevirapine in HIV infected adults (Monera Penduka et al., 2017).

A.3 OBJECTIVES List the major objectives/hypothesis, which have governed your choice of study design General objective

To determine the effect of Artemisia annua powder and Moringa oleifera on immunological and haematological response in patients on HAART.

Specific objectives

1. To determine effect of Artemisia annua in combination with Moringa oleifera on CD4 cell count in HIV patients on HAART.
2. To determine the effect of Artemisia annua with Moringa oleifera on viral load in patients on HAART.
3. To determine the effect of Artemisia annua with Moringa oleifera on full blood count and immunogloblins associated with HIV infections in HAART patients.
4. To determine the effect of Artemisia annua and Moringa oleifera on antiretroviral plasma drug level in patients on first line ART (UCG, 2016).
5. To determine the effect of Artemisia annua and Moringa oleifera on performance status and quality of life in HAART patients.
6. To profile any adverse effects of Artemisia annua and Moringa oleifera HIV patients on HAART.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is 18 years of age and above
2. Participant is HIV positive
3. Participant is on HAART first line for at least one year.
4. Participant is mentally sound
5. Participant is living within 60 km radius from the clinic and will be remaining within the radius of 60 km from the clinic during the study period

h) Participant has a CD4 count less than 350cells/µl i.)Participant has normal haematological and biochemical indices J) ability to use phone SMS messaging K) Participant has signed the informed consent form

Exclusion Criteria:

1. Participant is pregnant
2. Participant does not consent to study
3. Participant with opportunistic infection
4. Participants using other herbal medicines
5. Participant living outside the radius of 60 km from the clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-12-10 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
CD4 counts | Baseline, 6 and 12 months
  The primary outcome will be change in CD4 counts (absolute and relative) at 6 and 12 months in study participants following enrollment in the study.

SECONDARY OUTCOMES:
Viral load | Baseline, 6 and 12 months
  Viral load at baseline, 6 and 12 months from time of initiating herbal treatment with the above mentioned herbs.
Complete Blood Count | Baseline, 6 and 12 months
  Complete Blood Count at baseline, 6 and 12 months
Immunoglobins | Baseline, 6 and 12 months
  Immunoglobins (E, A, G) associated with HIV infections in HAART patients at baseline, 6 and 12 months
Antiretroviral plasma drug level | Baseline, one and two weeks
  Antiretroviral plasma drug level in HAART patients at baseline and after one and two weeks
Patients perceptions on mental and physical quality of life | Baseline, 6 and 12 months
  WHO Quality of life Tool-HIV
Liver function biomarkers | Baseline, 6 and 12 months
  Liver function biomarkers at baseline, six and twelve months
Side effects or adverse drug reactions | Baseline, 12 months
  Incidence of side effects or adverse drug reactions in the study participants over the study period
Renal function biomarkers | Baseline, 6 and 12 months
  Renal function biomarkers at baseline, six and twelve months

CONTACTS AND LOCATIONS:
Locations (1):
- Mbarara Regional Referral Hospital, Mbarara, SouthWestern, Uganda

IPD SHARING:
Plan to Share IPD: No
Participant lab results will be availed to the attending physician

REFERENCES:
- [Background] Alin MH, Ashton M, Kihamia CM, Mtey GJ, Bjorkman A. Clinical efficacy and pharmacokinetics of artemisinin monotherapy and in combination with mefloquine in patients with falciparum malaria. Br J Clin Pharmacol. 1996 Jun;41(6):587-92. doi: 10.1046/j.1365-2125.1996.35116.x. PMID 8799526
- [Background] Ashton M, Gordi T, Trinh NH, Nguyen VH, Nguyen DS, Nguyen TN, Dinh XH, Johansson M, Le DC. Artemisinin pharmacokinetics in healthy adults after 250, 500 and 1000 mg single oral doses. Biopharm Drug Dispos. 1998 May;19(4):245-50. doi: 10.1002/(sici)1099-081x(199805)19:43.0.co;2-z. PMID 9604124
- [Background] Zhao KC, Song ZY. [Pharmacokinetics of dihydroqinghaosu in human volunteers and comparison with qinghaosu]. Yao Xue Xue Bao. 1993;28(5):342-6. Chinese. PMID 8237378
- [Derived] Twinomujuni SS, Atukunda EC, Mukonzo JK, Nicholas M, Roelofsen F, Ogwang PE. Evaluation of the effects of Artemisia Annua L. and Moringa Oleifera Lam. on CD4 count and viral load among PLWH on ART at Mbarara Regional Referral Hospital: a double-blind randomized controlled clinical trial. AIDS Res Ther. 2024 Apr 16;21(1):22. doi: 10.1186/s12981-024-00609-4. PMID 38627722